CLINICAL TRIAL: NCT04792424
Title: No Monitoring of Post-filter Ionized Calcium in Regional Citrate Anticoagulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Nattachai Srisawat ,M.D., Director of Excellence Center for Critical Care Nephrology, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB.35/64
Record Dates: First submitted 2021-03-03; First posted 2021-03-11 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Regional Citrate Anticoagulation; Ionized Calcium; Continuous Renal Replacement Therapy
Keywords: Regional citrate anticoagulation; Ionized calcium; Continuous Renal Replacement Therapy
MeSH Terms: interventions — Vasoconstrictor Agents; Anti-Bacterial Agents; Dialysis; Continuous Renal Replacement Therapy

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: Masking of post-filter ionized calcium result in no-monitoring arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No monitoring of post filter ionized calcium (Experimental): Starting dialysis with continuous renal replacement therapy with regional citrate anticoagulation.
  Patients will receive standard treatments such as anti-bacterial agents, mechanical ventilator, vasopressors as appropriate.
  Citrate dose start at 4 mmol/L and no adjustment of citrate dose. Post-filter ionized calcium result will blind for physician.
  Other laboratory such as pre-filter ionized calcium, electrolyte, ABG, calcium, the ratio of total calcium to systemic ionized calcium will monitor every 8 hour.
  Interventions: Other: Regional citrate anticoagulation; Drug: Vasopressor; Drug: Antibiotic; Device: Dialysis with continuous renal replacement therapy
- Monitoring of post filter ionized calcium (Placebo Comparator): Starting dialysis with continuous renal replacement therapy with regional citrate anticoagulation.
  Patients will receive standard treatments such as anti-bacterial agents, mechanical ventilator, vasopressors as appropriate.
  Citrate dose start at 4 mmol/L with adjustment of citrate dose to acheive post-filter ionized calcium at 0.25-0.35 mmol/L.
  Other laboratory such as pre-filter ionized calcium, electrolyte, ABG, calcium, the ratio of total calcium to systemic ionized calcium will monitor every 8 hour.
  Interventions: Other: Regional citrate anticoagulation; Drug: Vasopressor; Drug: Antibiotic; Device: Dialysis with continuous renal replacement therapy

INTERVENTIONS:
Other: Regional citrate anticoagulation — Starting RCA 4 mmol/L (adjust the rate by BFR)
Drug: Vasopressor — Vasopressors such as Norepinephrine, dopamine, milrinone, dobutamine
Drug: Antibiotic — Antibacterial agents deemed appropriate by physicians in the ICU
Device: Dialysis with continuous renal replacement therapy — Prismaflex

SUMMARY:
Do no monitor of post-circuit ionized calcium affact the filter life time of continueous renal replacement therapy with regional citrate anticoagulation circuit? A randomized control trial

DETAILED DESCRIPTION:
Regional citrate anticoagulation is the gold standard of anticoagulation in patient receiving CRRT. In RCA circuit, there was a monitoring of pre-filter (systemic) ionized calcium and post-filter (circuit) ionized calcium. Pre-filter ionized calcium was monitored for observe the adverse effect of citrate such as hypocalcemia, citrate intoxication. However, post-filter ionized calcium was monitored for adjustment the citrate dose. We find many problem with frequently monitoring of post-ionized calcium such as confusion from markedly abnormal result, how to adjustment the citrate dose ,and increase workload for nurses. We hypothesis that if we can monitoring of post-filter ionized calcium?

ELIGIBILITY:
Inclusion Criteria:

* Age older than 18 years old and admission in an ICU
* Indication for CRRT
* regional citrate anticoagulation

Exclusion Criteria:

* Acute liver failure defined as AST or ALT > 5X UNL or TB/DB > 5X UNL or evidence of cirrhosis
* Severe persistent lactic acidosis (lactate persist > 8 mg/dL consecutively within 6 hours)
* Receiving heparin anticoagulation
* Severe alkalosis (pH>7.55) or acidosis (pH<7.1)
* History of renal allograft
* Known pregnancy
* Patient is moribund with expected death within 24 hr
* Deficiency of ionzed calcium (Cation < 0.8 mmol/L)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Filter lifetime in hours | 72 hours
  How long with filter with RCA

SECONDARY OUTCOMES:
Adverse event | 72 hours
  adverse event of RCA
Circuit downtime in hours | 72 hours
  Circuit downtime during CRRT with RCA
Cost per treatment in Baht | 72 hour
  Cost of CRRT include laboratory in Baht
Citrate accumulation | 72 hours
  Number of total calcium to ionized calcium ratio > 2.5
Efficacy of CRRT | 72 hours
  Seiving coefficient of urea and difference of prescribed dose of CRRT
Citrate dose | 72 hours
  Average citrate dose

OTHER OUTCOMES:
Change of SOFA scores | 72 hours
  Change of SOFA Scores (Use the worst value in 24 hour) from baseline to end of the study
Change of APACHE II score | 72 hours
  Change of APACHE II score (Use the worst value in 24 hour)from baseline to end of the study
Change of Hct | 72 hours
  Rate of Hct change from from baseline to end of the study
Change of electrolyte | 72 hours
  Rate of electrolyte change from baseline to end of the study

CONTACTS AND LOCATIONS:
Locations (1):
- Chulalongkorn university, Bangkok, Thailand

REFERENCES:
- [Derived] Thanapongsatorn P, Sinjira T, Kaewdoungtien P, Kusirisin P, Kulvichit W, Sirivongrangson P, Peerapornratana S, Lumlertgul N, Srisawat N. Standard versus no post-filter ionized calcium monitoring in regional citrate anticoagulation for continuous renal replacement therapy (NPC trial). Clin Kidney J. 2023 Mar 31;16(9):1469-1479. doi: 10.1093/ckj/sfad069. eCollection 2023 Sep. PMID 37664560